CLINICAL TRIAL: NCT02508948
Title: Current State of Endotracheal Intubation Among the Critically Ill and Exploring Risk Factors for Immediate Complications of Endotracheal Intubation: a Prospective, Observational Multi-center Study (HEMAIR)
Brief Title: Endotracheal Intubation Among the Critically Ill: HEMAIR Pilot Study
Acronym: HEMAIR
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Berkshire Medical Center (Other); Bridgeport Hospital (Other); Detroit Medical Center (Other); Geisinger Clinic (Other); Marshfield Clinic (Unknown); Memorial Medical Center (Other); Mercy Hospital (Unknown); University of North Carolina (Other); Johns Hopkins University (Other); University of Kentucky (Other); The Cleveland Clinic (Other); Wake Forest University Health Sciences (Other); Corpus Christi Medical Center (Unknown); University of Oklahoma (Other); Creighton University (Other); University of Southern California (Other); Essentia Health (Other)
Responsible Party: Principal Investigator, Nathan J. Smischney, PI, Mayo Clinic
Other Study IDs: 15-002328
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Tracheal Intubation
Keywords: airway management; critically ill; hemodynamic management; intubation; prospective study; risk factors
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
In order to examine the current endotracheal intubation practice among critically ill patients, a prospective observational multicenter study of adult critically ill patients was conducted from July 2015 to January 2017 involving 20 ICUs. In this study, the primary aim was to describe, through a prospective observational multicenter study, the current intubation practice of adult critically ill patients undergoing endotracheal intubations with a focus on deriving and validating a prediction model for both immediate airway and hemodynamic complications.

DETAILED DESCRIPTION:
Aim 1: To derive and validate a prediction model for difficult airway (three or more attempts at laryngoscopy to place an endotracheal tube and/or the need for another operator among the critically ill) [37].

Aim 2: To derive and validate a prediction model for hemodynamic compromise, i.e., post-intubation hypotension [defined as a decrease at any point in mean arterial pressure less than 65 mmHg; systolic blood pressure less than 80 mm Hg and/or a reduction in systolic blood pressure of 40% from baseline; or the initiation of, or increase in infusion dosage of, any vasopressor medication (bolus or infusion) during the 30 minute period following intubation] [38-39].

Aim3: To derive and validate a predication model for hypoxemia (decrease in pulse oximetry to oxygen saturation less than 88% during the procedure).

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Surgical and medical intensive care unit adult patients
* Adult patients requiring endotracheal intubation during the time period of study

Exclusion Criteria:

* Patient age < 18 years
* Endotracheal intubations performed outside the ICU (in the operating room, in and outside the hospital) are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to 20 participating medical/surgical/mixed ICUs who underwent endotracheal intubation.
Sampling Method: Probability Sample
Enrollment: 1288 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Hypoxemia in the 30 minutes following intubation | 30 minutes
Number of participants with hypotension in the 30 minutes following intubation | 30 minutes
Number of participants with unanticipated difficult airway | 10 minutes
  defined by 3 or more attempts or two operators

SECONDARY OUTCOMES:
Mechanical ventilation free days in-hospital | 28 days or in-hospital
Total days of ICU/hospital length of stay | 30 days or in-hospital
Number of participants with vital status (dead/alive) | 30 days or in-hospital
Number of participants with disposition to home, nursing home or long term care facility | 30 days or in-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Kashyap, MBBS, Study Director — Mayo Clinic
Locations (16):
- United States (16):
  - Mayo Clinic, Scottsdale, Scottsdale, Arizona
  - University of South California, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Bridgeport Hospital/Yale, Bridgeport, Connecticut
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - University of Kentucky, Lexington, Kentucky
  - Cynthia Callahan,Berkshire Medical Center, Pittsfield, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Mercy Hospital, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Health System, Danville, Pennsylvania
  - Corpus Christi Medical Center, Corpus Christi, Texas
  - Marshfield Clinic, Marshfield, Wisconsin
  - Arora Health Care, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smischney NJ, Surani SR, Montgomery A, Franco PM, Callahan C, Demiralp G, Tedja R, Lee S, Kumar SI, Khanna AK. Hypotension Prediction Score for Endotracheal Intubation in Critically Ill Patients: A Post Hoc Analysis of the HEMAIR Study. J Intensive Care Med. 2022 Nov;37(11):1467-1479. doi: 10.1177/08850666221085256. Epub 2022 Mar 4. PMID 35243921
- [Derived] Smischney NJ, Khanna AK, Brauer E, Morrow LE, Ofoma UR, Kaufman DA, Sen A, Venkata C, Morris P, Bansal V. Risk Factors for and Outcomes Associated With Peri-Intubation Hypoxemia: A Multicenter Prospective Cohort Study. J Intensive Care Med. 2021 Dec;36(12):1466-1474. doi: 10.1177/0885066620962445. Epub 2020 Oct 1. PMID 33000661
- [Derived] Smischney NJ, Kashyap R, Khanna AK, Brauer E, Morrow LE, Seisa MO, Schroeder DR, Diedrich DA, Montgomery A, Franco PM, Ofoma UR, Kaufman DA, Sen A, Callahan C, Venkata C, Demiralp G, Tedja R, Lee S, Geube M, Kumar SI, Morris P, Bansal V, Surani S; SCCM Discovery (Critical Care Research Network of Critical Care Medicine) HEMAIR Investigators Consortium. Risk factors for and prediction of post-intubation hypotension in critically ill adults: A multicenter prospective cohort study. PLoS One. 2020 Aug 31;15(8):e0233852. doi: 10.1371/journal.pone.0233852. eCollection 2020. PMID 32866219
- [Derived] Smischney N, Kashyap R, Seisa M, Schroeder D, Diedrich D. Endotracheal Intubation Among the Critically Ill: Protocol for a Multicenter, Observational, Prospective Study. JMIR Res Protoc. 2018 Dec 7;7(12):e11101. doi: 10.2196/11101. PMID 30530463
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials